CLINICAL TRIAL: NCT01841359
Title: Pramlintide (Symlin) for the Treatment of Hypoglycemia Following Gastric Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Joslin 08-34
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Results first posted 2022-05-26 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hypoglycemia; Evidence of Previous Gastric Surgery
Keywords: Hypoglycemia; Gastric bypass surgery
MeSH Terms: conditions — Hypoglycemia | interventions — pramlintide

STUDY DESIGN:
Intervention Model Description: Participants in this study were asked to complete 4 study visits.
  Arm/Phase 1: Baseline: Study V1 was a screening visit. Participants kept a 3-day log of food intake, blood glucose (8 per day), as well as any hypoglycemic symptoms. At V2, a baseline mixed meal tolerance test (MMTT) was performed. Glucose, hormonal responses, and satiety were assessed. Glucose and symptom logs were reviewed.
  Arm / Phase 2: Pramlintide treatment Pramlintide was prescribed at the end of visit 2 (following MMTT), with instructions for titration from minimal to maximal dose (15 to 120 µg). During treatment, the participants kept a record of all hypoglycemic symptoms and blood glucose measurements at those times.
  Study visit 3 occurred at week 4 of treatment and focused on evaluation of symptoms and side effects. Participants again completed a food and glucose diary for 3 days. During study visit 4 (week 8 of treatment), participants underwent a repeat MMTT.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline (No Intervention): Baseline Arm/Phase 1, is comprised of study visits 1 and 2. Visit 1: Screening visit. Eligible individuals who provided informed consent were asked to keep a 3-day log of food intake, blood glucose (8 per day), as well as any hypoglycemic symptoms, concurrent with a 3 day period of blinded (masked) continuous glucose monitoring device wear.
  Visit 2: a baseline mixed meal tolerance test was performed. Glucose, hormonal responses, and satiety were assessed. Glucose and symptom logs were reviewed.
- Pramlintide (Experimental): At the end of Visit 2 (following the baseline mixed meal tolerance test), pramlintide was prescribed, with instructions for titration from minimal to maximal dose (15 to 120 µg). During the treatment phase (8 weeks), the participants were asked to keep record of all hypoglycemic symptoms and blood glucose measurements..
  Visit 3: (week 4 of treatment) focused on evaluation of symptoms and side effects. Participants again completed a food and glucose diary for 3 days with concurrent wear of a blinded (masked) continuous glucose monitoring device.
  Visit 4: (week 8 of treatment), participants received a dose of pramlintide 15 minutes prior to undergoing a repeat mixed meal tolerance test. (the dose administered was the maximally tolerated dose of pramlintide used during the 8 week outpatient treatment phase).
  Interventions: Drug: Pramlintide

INTERVENTIONS:
Drug: Pramlintide — See description above (arm description).
  Other Names: Symlin
  Arms: Pramlintide

SUMMARY:
The purpose of this study is to determine whether pramlintide (Symlin) will help to reduce the frequency and severity of hypoglycemia in individuals who have had gastric bypass surgery.

DETAILED DESCRIPTION:
This study is an open-label short-term proof of concept study. The investigators will administer pramlintide to patients with severe post-prandial hypoglycemia following gastric bypass, in order to determine whether pramlintide is effective in reducing the frequency or severity of hypoglycemia. Pramlintide will be prescribed for 8 weeks. In order to assess the efficacy of pramlintide to prevent post-prandial hypoglycemia and hypoglycemic symptoms, the investigators will compare (a) blood glucose measurements and frequency of hypoglycemic symptoms, before and at the end of the drug intervention, using both capillary glucose monitoring and continuous glucose monitoring, and (b) glycemic, hormonal, and energetic responses to a three-hour mixed meal tolerance test.

The study will utilize an open label design to evaluate the efficacy of pramlintide in patients who have had gastric bypass and have severe postprandial hypoglycemia. The study will not be randomized or blinded. The investigators will recruit 26 participants from Joslin Diabetes Center.

Briefly, participants in this study will be asked to complete 4 study visits. The first visit will be for screening. They will then be asked to keep a 3-day log in which they record food intake (including estimated portion sizes), blood glucoses eight times daily, as well as any hypoglycemic symptoms, before they initiate treatment. Concurrently participants will wear a professional (blinded) continuous glucose monitoring (CGM) device for 3 days. At a second study visit, they will undergo a mixed meal tolerance test, which will serve as a baseline evaluation. Patterns of (a) glucose excursions (initial postprandial peak, subsequent postprandial fall and potential hypoglycemia), and (b) hormonal responses (insulin, C-peptide, glucagon, incretins) will be assessed. At the end of the mixed meal, satiety will be assessed using a visual analog scale. Baseline hypoglycemia frequency and severity will be assessed by reviewing patient glucose and hypoglycemia symptom log recorded prior to the visit.

At the completion of visit 2, pramlintide will be prescribed, with instructions for titration of the drug from minimal to maximal dose (see titration schedule below) to help reduce the incidence of side effects. During the treatment period, the participants will keep a record of all hypoglycemic symptoms and blood glucose measurements at those times.

There will be one follow-up visit (visit 3) in the middle of the treatment period for evaluation of symptoms and tolerance of medication. During the last (eighth) week of treatment, for comparison with pre-treatment glycemia, participants will again complete a food diary, and measure and record blood glucoses eight times daily for 3 days, while also wearing a professional (blinded) CGM. During that final week of the study, participants will also come to a fourth study visit, during which they will undergo a repeat mixed meal tolerance test, receiving a dose of pramlintide prior to the start of the mixed meal, for comparison with the pre-treatment (baseline) results.

ELIGIBILITY:
Inclusion Criteria:

* severe hypoglycemic episodes post-gastric bypass surgery
* normal fasting glucose
* age 21 to 65
* hypoglycemia must not have responded to dietary intervention (low glycemic index, controlled carbohydrate portions) and a trial of acarbose therapy at the maximally tolerated dose

Exclusion Criteria:

* Hypoglycemia in the fasting state (greater than 12 hours fast)
* History of preoperative diabetes mellitus
* Use of medications that affect gastrointestinal motility (e.g., cisapride, metoclopramide)
* Impaired renal function (creatinine clearance < 20 ml/min or on dialysis
* Hepatic disease (defined as liver enzymes > 2 times upper normal limit for alanine transaminase (ALT) and aspartate aminotransferase (AST))
* Blood donation for 2 months prior to the study.
* Severe hypoglycemic unawareness, as defined by inability to recognize adrenergic or neuroglycopenic symptoms of hypoglycemia despite detailed education

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Patti ME, Goldfine AB. Hypoglycaemia following gastric bypass surgery--diabetes remission in the extreme? Diabetologia. 2010 Nov;53(11):2276-9. doi: 10.1007/s00125-010-1884-8. Epub 2010 Aug 21. PMID 20730413
- [Background] Goldfine AB, Mun EC, Devine E, Bernier R, Baz-Hecht M, Jones DB, Schneider BE, Holst JJ, Patti ME. Patients with neuroglycopenia after gastric bypass surgery have exaggerated incretin and insulin secretory responses to a mixed meal. J Clin Endocrinol Metab. 2007 Dec;92(12):4678-85. doi: 10.1210/jc.2007-0918. Epub 2007 Sep 25. PMID 17895322
- [Background] Patti ME, McMahon G, Mun EC, Bitton A, Holst JJ, Goldsmith J, Hanto DW, Callery M, Arky R, Nose V, Bonner-Weir S, Goldfine AB. Severe hypoglycaemia post-gastric bypass requiring partial pancreatectomy: evidence for inappropriate insulin secretion and pancreatic islet hyperplasia. Diabetologia. 2005 Nov;48(11):2236-40. doi: 10.1007/s00125-005-1933-x. Epub 2005 Sep 30. PMID 16195867
- [Background] Goldfine AB, Mun E, Patti ME. Hyperinsulinemic hypoglycemia following gastric bypass surgery for obesity. Current Opinion in Endocrinology and Diabetes 13: 419-24, 2006.
- [Background] Sheehan A, Goldfine A, Bajwa M, Wolfs D, Kozuka C, Piper J, Fowler K, Patti ME. Pramlintide for post-bariatric hypoglycaemia. Diabetes Obes Metab. 2022 Jun;24(6):1021-1028. doi: 10.1111/dom.14665. Epub 2022 Mar 9. PMID 35137513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with post-bariatric hypoglycemia (PBH) following gastric bypass were recruited from outpatient clinics at Joslin Diabetes Center, Boston, Massachusetts for an open label study of pramlintide efficacy over 8 weeks.
Groups:
- Pramlintide (Symlin): Participants in this study were asked to complete 4 study visits. Study visit 1 was a screening visit. Eligible individuals who provided informed consent were asked to keep a 3-day log of food intake, blood glucose (8 per day), as well as any hypoglycemic symptoms. At study visit 2, a baseline mixed meal tolerance test was performed. Glucose, hormonal responses, and satiety were assessed. Glucose and symptom log was reviewed. Pramlintide was prescribed, with instructions for titration from minimal to maximal dose (15 to 120 µg). During treatment, the participants kept a record of all hypoglycemic symptoms and blood glucose measurements at those times.
  Study visit 3 occured at week 4 of treatment and focused on evaluation of symptoms and side effects. Participants again completed a food and glucose diary for 3 days. During study visit 4 (week 8 of treatment), participants underwent a repeat mixed meal tolerance test.
  Pramlintide: See description above (arm description).
Period: Overall Study
Arm/Group | Pramlintide (Symlin)
Started | 22
Completed | 14
Not Completed | 8
Not completed — Underwent reversal of Roux-en-Y gastric bypass (RYGB) | 2
Not completed — Concommitant medical issues | 2
Not completed — Adverse Event | 3
Not completed — Did not receive study drug at visit 4 prior to mixed meal testing | 1

BASELINE CHARACTERISTICS:
Population: Analysis is based upon 14 participants who completed the protocol.
Groups:
- Pramlintide (Symlin): Participants in this study completed 4 study visits. Study visit 1 was a screening visit. Participants kept a 3-day log of food intake, blood glucose (8 per day), as well as any hypoglycemic symptoms. At study visit 2, a baseline mixed meal tolerance test were performed. Glucose, hormonal responses, and satiety were assessed. Glucose and symptom log was reviewed. Pramlintide was prescribed, with instructions for titration from minimal to maximal dose (15 to 120 µg). During treatment, the participants kept a record of all hypoglycemic symptoms and blood glucose measurements at those times.
  Study visit 3 occurred at week 4 of treatment and focused on evaluation of symptoms and side effects. Participants again completed a food and glucose diary for 3 days. During study visit 4 (week 8 of treatment), participants underwent a repeat mixed meal tolerance test.
  Pramlintide: See description above (arm description).
Arm/Group | Pramlintide (Symlin)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 14
Pre-operative BMI [Mean (Standard Deviation); unit: kg/m^2] | 46.8 (6.2)
Current BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (4.3)
Onset of hypoglycemia (years since) surgery [Mean (Standard Deviation); unit: years] | 2.9 (2.9)
Time Since RYGB (years) [Mean (Standard Deviation); unit: years] | 6.2 (2.7)
Preoperative history of diabetes mellitus (DM) or gestational DM [Count of Participants; unit: Participants] | 3
Family history of DM in first-degree relative [Count of Participants; unit: Participants] | 6
Possible hypoglycemia symptoms present preoperatively (self-report) [Count of Participants; unit: Participants] | 2
Hypoglycemia frequency (self-report) - Daily or more [Count of Participants; unit: Participants] | 1
Hypoglycemia frequency (self-report) - Weekly or more (but not daily) [Count of Participants; unit: Participants] | 7
Hypoglycemia frequency (self-report) - Monthly or more (but not weekly) [Count of Participants; unit: Participants] | 1
Systolic Blood Pressure Supine [Mean (Standard Deviation); unit: mmHg] | 119.1 (12.5)
Diastolic Blood Pressure Supine [Mean (Standard Deviation); unit: mmHg] | 67.8 (10.3)
Cholesterol (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 169.6 (18.2)
Triglycerides (mg/dl) [Mean (Standard Deviation); unit: mg/dL] | 75.2 (20.2)
HDL (mg/dl) [Mean (Standard Deviation); unit: mg/dL] | 64.6 (10.1)
Current therapy with acarbose [Count of Participants; unit: Participants] | 8
Current therapy with diazoxide [Count of Participants; unit: Participants] | 0
Current therapy with octreotide [Count of Participants; unit: Participants] | 1
Current therapy - medical nutrition therapy alone [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose Levels in Response to Mixed Meal Testing - Area Under the Curve for Plasma Glucose
Description: Baseline and post-treatment with pramlintide mixed meal testing plasma glucose values, area under the curve (AUC), calculated with the trapezoidal method.
  Plasma glucose was measured at timepoints (minutes): -5 (baseline), 10 minutes, 20 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes.
Time Frame: Levels assessed on the two days of mixed meal testing: the first occurring at baseline; and the second following 8 weeks of treatment with pramlintide.
Population: Analysis was for the 14 participants who completed all study visits.
Measure: Geometric Mean (Standard Deviation); unit: mg*min/dL
Groups:
- Baseline (Prior to Pramlintide Treatment) Mixed Meal #1: Mixed meal #1 performed prior to initiation of pramlintide treatment.
- Pramlintide - Mixed Meal #2: Mixed meal #2 performed after 1 dose of pramlintide given 15 minutes prior to the mixed meal, at maximum tolerated dose achieved during the outpatient stage.
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
mg*min/dL | 2828 (3255) | 2893 (2770)
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.90, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Continuous Glucose Monitoring Maximum Sensor Glucose Values Prior to (Baseline) and During Pramlintide Therapy.
Time Frame: During 8 week period of participation, V1-V2 (baseline CGM data over 3 days); V3-V4 (CGM data during treatment with three times per day (TID) pramlintide over 3 days)
Population: Analysis was for the participants with available CGM data who completed all study visits in this sequential design. Note that the number of participants analyzed for CGM related outcomes differs from the number of participants analyzed in the other outcomes due to incomplete CGM data.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Baseline (Prior to Treatment With Pramlintide) CGM #1: Stage 1 of sequential design. Participant CGM data at baseline, prior to initiation of treatment with pramlintide TID.
- Pramlintide CGM #2: Stage 2 of sequential design. Participant CGM data during treatment with pramlintide TID.
Arm/Group | Baseline (Prior to Treatment With Pramlintide) CGM #1 | Pramlintide CGM #2
Number analyzed (Participants) | 13 | 10
mg/dL | 172 (50.98) | 188 (43.6)
Statistical Analysis 1: Comparison: Baseline (Prior to Treatment With Pramlintide) CGM #1 vs Pramlintide CGM #2; Test type: Other; p = 0.08, t-test, 2 sided

3. Secondary Outcome: Continuous Glucose Monitoring Minimum Sensor Glucose Prior to (Baseline) and During Pramlintide Therapy.
Time Frame: During 8 week period of participation, V1-V2 (baseline CGM data over 3 days); V3-V4 (CGM data during treatment with TID pramlintide over 3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline (Prior to Treatment With Pramlintide) CGM #1 | Pramlintide CGM #2
Number analyzed (Participants) | 13 | 10
mg/dL | 54 (14.68) | 56.6 (11.44)
Statistical Analysis 1: Comparison: Baseline (Prior to Treatment With Pramlintide) CGM #1 vs Pramlintide CGM #2; Test type: Other; p = 0.20492, t-test, 2 sided

4. Secondary Outcome: Hypoglycemia - Percentage of Time Sensor Glucose Levels < 70 mg/dL Prior to (Baseline) and During Pramlintide Therapy.
Description: Assessment of clinical response to pramlintide treatment, as indicated by paired comparison of the frequency of glucose values under 70 mg/dl (expressed as percentage of time) assessed by continuous glucose monitoring.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent time sensor glucose less than 70
Arm/Group | Baseline (Prior to Treatment With Pramlintide) CGM #1 | Pramlintide CGM #2
Number analyzed (Participants) | 13 | 10
percent time sensor glucose less than 70 | 8.85 (9.23) | 5.60 (5.32)
Statistical Analysis 1: Comparison: Baseline (Prior to Treatment With Pramlintide) CGM #1 vs Pramlintide CGM #2; Test type: Other; p = 0.2655, t-test, 2 sided

5. Secondary Outcome: Plasma Insulin Levels in Response to Mixed Meal Testing - Area Under the Curve for Plasma Insulin
Description: Pre- and post-treatment mixed meal testing plasma insulin levels area under the curve (AUC) was calculated with the trapezoidal method.
  Plasma insulin was measured at timepoints (minutes): -5 (baseline), 10 minutes, 20 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes.
Time Frame: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: uIU*min/mL
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
uIU*min/mL | 3393 (2155) | 3501 (2683)
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.64, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Satiety Score During Mixed Meal Testing at 120 Minutes
Description: Satiety was analyzed using a visual analogue scale (1, very hungry to 10, not hungry), administered 120 minutes following ingestion of mixed meal.
Time Frame: Levels assessed on the two days of mixed meal testing at the 120 min time point: the first occurring at baseline (prior to treatment with pramlintide), and the second following 8 weeks of treatment with pramlintide.
Measure: Mean (Standard Deviation); unit: satiety score
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
satiety score | 4.57 (3.05) | 5.43 (2.51)
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.597, t-test, 2 sided

7. Secondary Outcome: Dumping Score During Mixed Meal Testing at Baseline and During Treatment With Pramlintide
Description: Dumping score was calculated using changes in pulse and hematocrit. Higher scores indicate more severe dumping. Scores ranged from -196 to 186.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: dumping score
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
dumping score | 28.89 (101.81) | 72.04 (70.93)
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.37, t-test, 2 sided

8. Secondary Outcome: Number of Days With Minimum Sensor Glucose < 54 mg/dL as Measured by Continuous Glucose Monitoring.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Baseline (Prior to Treatment With Pramlintide) CGM #1 | Pramlintide CGM #2
Number analyzed (Participants) | 13 | 10
days | 1.31 (1.49) | 0.56 (0.73)
Statistical Analysis 1: Comparison: Baseline (Prior to Treatment With Pramlintide) CGM #1 vs Pramlintide CGM #2; Test type: Other; p = 0.14, t-test, 2 sided

9. Secondary Outcome: Nadir Plasma Glucose Levels During Mixed Meal Testing at Baseline and During Treatment With Pramlintide
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
mg/dL | 67.18 (17.14) | 69.9 (14.8)
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.412, t-test, 2 sided

10. Secondary Outcome: Time to Nadir Plasma Glucose During Mixed Meal Testing at Baseline and During Treatment With Pramlintide
Time Frame: Assessed on the two days of mixed meal testing: the first occurring at baseline; and the second following 8 weeks of treatment with pramlintide.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
minutes | 64.29 (40.52) | 66.43 (48.77)
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.890, t-test, 2 sided

11. Secondary Outcome: Number of Participants Requiring Rescue Treatment for Severe Hypoglycemia During Mixed Meal Testing (Visit 2 Baseline vs. Visit 4 Post-pramlintide Dosing)
Time Frame: as for outcome 10
Measure: Number; unit: number of participants
Arm/Group | Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 | Pramlintide - Mixed Meal #2
Number analyzed (Participants) | 14 | 14
number of participants | 6 | 4
Statistical Analysis 1: Comparison: Baseline (Prior to Pramlintide Treatment) Mixed Meal #1 vs Pramlintide - Mixed Meal #2; Test type: Other; p = 0.69, Fisher Exact

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data was collected during their 8 week period of participation. Overall, the participant data was collected from April 2014 through May 2016.
Arm/Group | Pramlintide (Symlin)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramlintide (Symlin) (N=22)
Dehydration (r/t diarrhea) (General disorders) | 1 (1) — Not related to study drug / procedures (onset was prior to study drug initiation). Pt was hospitalized 24 hrs. Resolved.
Diarrhea (assoc. with dehydration requiring hospitalization) (Gastrointestinal disorders) | 1 (1) — Associated with dehydration. Not related to study drug / procedures (onset was prior to study drug initiation). Pt was hospitalized 24 hrs. Resolved.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramlintide (Symlin) (N=22)
Hypoglycemia (Endocrine disorders) | 4 — Baseline (pre-study drug start) hypoglycemia (n=2) During study drug treatment hypoglycemia (n=2)
Hyperglycemia (Endocrine disorders) | 1 — Capillary glucose 450. Related to post-bariatric surgery status (rapid absorption / high peak of glucose levels).
Elevated liver enzymes (Hepatobiliary disorders) | 1 — Alcohol use acknowledged by participant, started on Campral since 10/18/14. Recovered / resolved.
Nausea (General disorders) | 3 — Possibly related to study drug. Pramlintide doses reduced (n=2). Nausea resolved or improved to baseline level of pre-existing nausea.
Altered taste (during treatment with study drug) (General disorders) | 1 — Related.
Ethanol abuse / intoxication (Psychiatric disorders) | 1 — Withdrawn from study, referred for support (AA, detox, alcohol detox specialist).
Trembling (General disorders) | 1 — Resolved. Related to treatment. Withdrawn from study due to multiple symptoms related to treatment.
Diarrhea (with urgency and incontinence) (Gastrointestinal disorders) | 1 — Resolved.
Auditory hallucinations (Psychiatric disorders) | 1 — Resolved. Related to treatment. Withdrawn from study due to multiple symptoms related to treatment.
Cold feeling behind eyes. (General disorders) | 1 — Resolved. Related to treatment. Withdrawn from study due to multiple symptoms related to treatment.
Nightmares (General disorders) | 1 — Resolved. Related to treatment. Withdrawn from study due to multiple symptoms related to treatment.
Increase in baseline anxiety. (Psychiatric disorders) | 1 — Withdrawn from study due to multiple symptoms related to treatment.
Symptoms of a urinary tract infection (UTI) (CVA tenderness w/ dysuria) (Renal and urinary disorders) | 1 — No abnormal labs at V1/V2. U/A was negative for a urinary tract infection. Recovered without sequelae.
Cholecystitis (prior to treatment with study drug) (Hepatobiliary disorders) | 1 — Not related. Preexisting condition identified during screening process, patient not enrolled in study at that time. Not related recovered without sequelae.
Sinus infection (Visit 4, following treatment with study drug) (Respiratory, thoracic and mediastinal disorders) | 1 — Not related. Recovered without sequelae.
Weight loss (during study drug treatment) (General disorders) | 1 — Possibly related. 6.6 lbs in 6 weeks. Related. Study drug dose decreased from 60 mcg to 30 mcg. Recovered without sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes